CLINICAL TRIAL: NCT00039819
Title: Plasticity of Reciprocal Inhibition
Brief Title: Nerve Stimulation to Modify a Spinal Reflex
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020228; 02-N-0228
Record Dates: First submitted 2002-06-11; First posted 2002-06-12 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-05

CONDITIONS: Healthy
Keywords: Spinal Cord; Sensory Stimulation; Locomotion; Magnetic Stimulation; Reflexes; Healthy Volunteer; HV; Normal Control

SUMMARY:
This study will determine whether stimulating the nerves or the brain can modify the spinal reflex that controls the muscles that flex and extend the ankle. Training spinal nerve networks with sensory input may provide a way of re-establishing movements, such as walking, in patients with spinal injury.

Healthy normal volunteers with no history of peripheral neuropathy or radiculopathy, ankle contractures or tendon surgery may be eligible for this study. Participants will undergo three stimulation procedures, each in a different session, to measure leg muscle reflexes. The procedures are:

* Reflex testing - Metal electrodes are taped to the skin over the leg muscles. A small electrical pulse is delivered through the electrodes to stimulate two nerves to the muscles. This evokes a reflex between the ankle flexor and extensor muscles. The responses to several dozen stimuli are averaged.
* Nerve stimulation - The nerve to the muscle that flexes the leg is electrically stimulated near the knee through electrodes taped to the skin. The strength of the stimulus is adjusted to produce little or no muscle movement. The stimulation is repeated every few seconds for 45 minutes.
* Transcranial magnetic stimulation - An insulated wire coil is placed on the subject's scalp. A brief electrical current passes through the coil, creating a magnetic pulse that travels through the scalp and skull and causes small electrical currents in the outer part of the brain. There may be twitching in the muscles of the arm or leg. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions to help determine the best position for the coil over the part of the brain that controls the leg. The leg is then stimulated once every 10 seconds, combined with nerve stimulation every 1 to 2 seconds.

DETAILED DESCRIPTION:
Training of spinal interneuronal networks may offer a means for re-establishing movements such as locomotion in patients with spinal injury. Sensory feedback in the pattern which results from the leg movement is hypothesized to be the critical component for training spinal networks. This protocol will address the basic assumption underlying such training: can a specific pattern of sensory input modify the strength of a spinal cord circuit? We will test whether peripheral nerve stimulation can modify the strength of the spinal reflex mediating reciprocal inhibition between ankle flexor and extensor muscles in normal subjects, comparing patterned and unpatterned stimulation.

ELIGIBILITY:
INCLUSION CRITERIA:

Healthy adult volunteers willing to participate

EXCLUSION CRITERIA:

History of peripheral neuropathy or radiculopathy

Implanted devices, including pacemakers, pumps, and defibrillators

Ankle contractures or tendon surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2002-06; Study Completion 2003-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Burke RE. The central pattern generator for locomotion in mammals. Adv Neurol. 2001;87:11-24. No abstract available. PMID 11347213
- [Background] Wirz M, Colombo G, Dietz V. Long term effects of locomotor training in spinal humans. J Neurol Neurosurg Psychiatry. 2001 Jul;71(1):93-6. doi: 10.1136/jnnp.71.1.93. PMID 11413270
- [Background] Rossignol S. Locomotion and its recovery after spinal injury. Curr Opin Neurobiol. 2000 Dec;10(6):708-16. doi: 10.1016/s0959-4388(00)00151-3. PMID 11240279